CLINICAL TRIAL: NCT06262035
Title: Transcriptome, Proteome and Microbiome Profile in Periodontal and Peri-implant Diseases
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Tülay Yucel Lindberg, Associate Professor, Karolinska Institutet
Other Study IDs: 2023-02987-01
Record Dates: First submitted 2024-01-25; First posted 2024-02-15 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Peri-implantitis; Periodontitis
Keywords: Peri-implantitis; Periodontitis
MeSH Terms: conditions — Peri-Implantitis; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Gingival crevicular fluid Peri-implant crevicular fluid Soft tissue biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Periodontitis and Peri-implantitis — Defined periodontitis at ≤ 2 non-adjacent teeth AND Defined peri-implantitis at ≤ 1 implant, in function of at least 1 year.

SUMMARY:
1. To investigate the transcriptomic profile of periodontitis and peri-implantitis. Patients with defined periodontitis, at two non-adjacent teeth and peri-implantitis at ≥ one implant in function of ≥ one year, will be included to investigate the gene expression profile in tissue affected by periodontitis and peri-implantitis. Subjects will undergo a full-mouth examination performed by a calibrated examiner, including assessment of caries, bone abnormalities and infections according to intraoral x-ray, plaque index and pocket probing depth, suppuration, bleeding on probing, alveolar bone loss, and the number of teeth. During surgical intervention, tissue biopsies (two specimens per site) will be collected by a periodontist from site with ongoing periodontitis and site from ongoing peri-implantitis.
2. To study the microbiome and biomarker profile associated with periodontitis and peri- implantitis. Patients with defined periodontitis, at two non-adjacent teeth and peri-implantitis at ≥ one implant in function of ≥ one year, will be included in this study to determine the bacteria composition, cytokine profile and inflammatory biomarkers profile. Subjects will undergo a full-mouth examination performed by a calibrated examiner, including assessment of caries, bone abnormalities and infections according to intraoral x-ray, plaque index and pocket probing depth, suppuration, bleeding on probing, alveolar bone loss, and number of teeth. Peri-implant crevicular fluid (PICF), gingival crevicular fluid (GCF), saliva and submucosal/subgingival plaque will be collected.The presence and composition of periodontal and peri-implant plaque samples are investigated.

ELIGIBILITY:
Inclusion Criteria:

≥18 years of age Defined periodontitis at two non-adjacent teeth Defined peri-implantitis at ≥1 implant Signed informed consent

Exclusion Criteria:

Surgical intervention of periodontitis and/or peri-implantitis during last 6 months.

Local or systemic use of antibiotics during last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with periodontitis and peri-implantitis, referred from a general clinic in Stockholm County to a periodontist.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Protein levels in peri-implantitis and periodontitis | Through study completion, an average of 1 years
  To measure protein levels in gingival crevicular fluid and in peri-implant crevicular fluid.
Microbiome composition in peri-implantitis and periodontitis using 16S-rRNA sequencing method. | Through study completion, an average of 1 years
  The microbiome composition will be analyzed in samples of subgingival/submucosal plaque using 16S-rRNA sequencing method.
Gene expression profile in peri-implantitis and periodontitis. | Through study completion, an average of 1 years
  Soft tissue specimens will be studied in regards of gene expression levels using RNA sequencing method (Ilumina). The mRNA expression of candidate genes will be studied at protein level using immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Tülay Lindberg, Ass.prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Aqua Dental Specialistklinik, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No